CLINICAL TRIAL: NCT00566332
Title: Randomized Trial Comparing the Efficacy of Chlorambucil to Fludarabine in Patients With Advanced Waldenström Macroglobulinemia,Lymphoplasmacytic Lymphoma or Splenic Marginal Zone Lymphoma
Brief Title: Trial Comparing Chlorambucil to Fludarabine in Patients With Advanced Waldenström Macroglobulinemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: French Study Group on Chronic Lymphoid Leukemia (Network)
Collaborators: Lymphoma Study Association (Other); French Innovative Leukemia Organisation (Other); Département de Biostatistiques et Informatique Médicale DBIM (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WM1
Record Dates: First submitted 2007-11-30; First posted 2007-12-03 (Estimated); Last update posted 2015-08-19 (Estimated); Status verified 2015-08

CONDITIONS: Waldenström Macroglobulinemia; Lymphoplasmacytic Lymphoma; Splenic Marginal Zone Lymphoma
Keywords: Waldenström Macroglobulinemia; Lymphoplasmacytic lymphoma; Splenic Marginal Zone Lymphoma; Fludarabine; Chlorambucil
MeSH Terms: conditions — Waldenstrom Macroglobulinemia; Lymphoma, B-Cell, Marginal Zone | interventions — Chlorambucil; fludarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Chlorambucil 8mg/m² (6 mg/m² if patient aged more than 75 years old) 10 days every 28 days during 12 months
  Interventions: Drug: Chlorambucil
- 2 (Active Comparator): Fludarabine
  Interventions: Drug: Fludarabine

INTERVENTIONS:
Drug: Chlorambucil — Chlorambucil 8 mg/m² (6 mg/m² if patient aged more than 75 years old) 10 days every 28 days during 12 months By oral route
  Arms: 1
Drug: Fludarabine — Fludarabine 40 mg/m² (30 mg/m² if patient aged more than 75 years old) 5 days every 28 days during 6 cycles By oral route
  Arms: 2

SUMMARY:
Waldenström's macroglobulinaemia (WM) is a lymphoproliferative disorder characterized by a monoclonal IgM paraprotein and morphological evidence of lymphoplasmacytic lymphoma: the cells are IgM+, IgD+, CD19+ and CD20+ but usually CD5-, CD10- and CD23-. The treatment efficacy is difficult to assess because of the lack of clear diagnostic criteria , good response criteria, and of randomized trials.

The actual treatment is Chlorambucil, an alkylating agent. A purine analogue such as Fludarabine has proven its efficacy on 30 % to 80 % as first line therapy

This study is a phase II b open, prospective, international multicenter trial (England, Dr Johnson, Dr Catovsky, Australia: Dr Seymour) promoted by the French Cooperative Group on Chronic Lymphoid Leukemia in untreated WM, or closely related disorders ( Lymphoplasmacytic lymphoma or splenic marginal zone lymphoma). 366 patients must be included, among them 180 patients in France. Patients will be stratified according to the lymphoproliferative disorder.

The patients will receive Chlorambucil by oral route for 10 days every 28 days (12 cycles) (8 MG/M², 6 MG/M² if patient is more than 75 years old) or Fludarabine by oral route for 5 days every 28 days (6 cycles) (40MG/M², 30 MG/M² if patient is more than 75 years old).

The primary objective is to compare the efficacy (response rate) of Chlorambucil to Fludarabine in previously untreated patients. The secondary objectives are the duration of response, the improvement of hematological parameters, the toxicity, the quality of life, the event free survival and the overall survival.

ELIGIBILITY:
Inclusion Criteria:

Established diagnosis of Waldenström macroglobulinemia (the 2nd Workshop on Waldenstrom's macroglobulinemia) or Lymphoplasmacytic lymphoma or Splenic Marginal Zone Lymphoma, needing a treatment

* Life expectancy > 6 months
* Creatinine < 200 µmol/l
* SGPT and SGOT < 2x ULN
* A negative direct Coombs test
* Written informed consent

Exclusion Criteria:

* Past chemotherapy/radiotherapy/immunotherapy prior to the study for Waldenström macroglobulinemia
* Previous malignancy less than 5 years ago except carcinoma in situ of the cervix and non-melanoma skin cancer
* Positive HIV serology
* Active Hepatitis B or C
* Lactation/pregnancy
* Impossible good compliance with the study protocol
* Active infection not controlled
* Psychological condition hampering understanding of the study
* Transformation into large B cell lymphoma
* Peripheral neuropathy > grade II

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 414 (Actual)
Dates: Start 2001-06; Primary Completion 2009-09 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Patient overall response | At the end of treatment whether 6 or 12 months

SECONDARY OUTCOMES:
Biological study | Whether 6 or 12 months
Quality of life | Whether 6 or 12 months
Response duration | 60 months
Treatment toxicity | 60 months
Event free survival | 60 months
Overall survival | 60 months

CONTACTS AND LOCATIONS:
Overall Officials: Véronique LEBLOND, Professor, Principal Investigator — French Study Group on Chronic Lymphoid Leukemia
Locations (1):
- Hôpital La Pitié-Salpêtrière. 47-83 Bd de l'hôpital, Paris, France

REFERENCES:
- [Derived] Leblond V, Johnson S, Chevret S, Copplestone A, Rule S, Tournilhac O, Seymour JF, Patmore RD, Wright D, Morel P, Dilhuydy MS, Willoughby S, Dartigeas C, Malphettes M, Royer B, Ewings M, Pratt G, Lejeune J, Nguyen-Khac F, Choquet S, Owen RG. Results of a randomized trial of chlorambucil versus fludarabine for patients with untreated Waldenstrom macroglobulinemia, marginal zone lymphoma, or lymphoplasmacytic lymphoma. J Clin Oncol. 2013 Jan 20;31(3):301-7. doi: 10.1200/JCO.2012.44.7920. Epub 2012 Dec 10. PMID 23233721
- [Derived] Nguyen-Khac F, Lambert J, Chapiro E, Grelier A, Mould S, Barin C, Daudignon A, Gachard N, Struski S, Henry C, Penther D, Mossafa H, Andrieux J, Eclache V, Bilhou-Nabera C, Luquet I, Terre C, Baranger L, Mugneret F, Chiesa J, Mozziconacci MJ, Callet-Bauchu E, Veronese L, Blons H, Owen R, Lejeune J, Chevret S, Merle-Beral H, Leblondon V; Groupe Francais d'Etude de la Leucemie Lymphoide Chronique et Maladie de Waldenstrom (GFCLL/MW); Groupe Ouest-Est d'etude des Leucemie Aigues et Autres Maladies du Sang (GOELAMS); Groupe d'Etude des Lymphomes de l'Adulte (GELA). Chromosomal aberrations and their prognostic value in a series of 174 untreated patients with Waldenstrom's macroglobulinemia. Haematologica. 2013 Apr;98(4):649-54. doi: 10.3324/haematol.2012.070458. Epub 2012 Oct 12. PMID 23065509